CLINICAL TRIAL: NCT05913323
Title: Measuring Lung Mechanics in Patients with Chronic Obstructive Pulmonary Disease (COPD) Using the Rapid Expiratory Occlusion Method (REOM) Handheld Portable Oscillometer: a Cross-Sectional Study.
Brief Title: Measuring Lung Mechanics in Patients with COPD Using the REOM Handheld Portable Device
Status: Completed | Type: Observational
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: McGill University (Other); Thorasys Thoracic Medical Systems Inc. (Industry)
Responsible Party: Principal Investigator, Bryan Ross, Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: 2023-9001
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Copd
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- COPD sub-group: GOLD 1 COPD: A secondary objective of the study is to investigate the discriminative capacity of the parameters obtained from the REOM to distinguish between 'mild' and 'very severe' COPD.
  Thus, there will be a 'mild' (GOLD 1) COPD sub-group.
  Interventions: Device: Rapid Expiratory Occlusion Monitor (REOM); Diagnostic Test: Standard oscillometry; Diagnostic Test: Standard pulmonary function test
- COPD sub-group: GOLD 4 COPD: A secondary objective of the study is to investigate the discriminative capacity of the parameters obtained from the REOM to distinguish between 'mild' and 'very severe' COPD.
  Thus, there will be a 'very severe' (GOLD 4) COPD sub-group.
  Interventions: Device: Rapid Expiratory Occlusion Monitor (REOM); Diagnostic Test: Standard oscillometry; Diagnostic Test: Standard pulmonary function test

INTERVENTIONS:
Device: Rapid Expiratory Occlusion Monitor (REOM) — Device for which Health Canada approval (ITA Authorization) has been obtained for use in the present study.
Diagnostic Test: Standard oscillometry — tremoflo device-100, Thorasys Thoracic Medical Systems Inc., Montreal, Canada
Diagnostic Test: Standard pulmonary function test — Standard-of-care respiratory test.

SUMMARY:
The purpose the study is to determine the agreement between the information obtained about lung mechanics (lung function) from the Rapid Expiratory Occlusion Monitor (REOM) handheld portable device with that obtained by conventional oscillometry as well as by pulmonary function testing (PFT), in patients with both 'mild' as well as 'very severe' forms of chronic obstructive pulmonary disease (COPD). This study also intends to study the user experience with this handheld portable device.

DETAILED DESCRIPTION:
The primary objective of this cross-sectional study is to determine the concordance and agreement between the parameters obtained from the REOM, Reo1 and Reo2, and the conventional resistance parameters obtained by the tremoflo oscillometer device (R19 and R5, respectively) in adults with COPD confirmed by diagnostic pulmonary function testing (PFT).

The secondary objectives are:

1. To investigate the discriminative capacity of the parameters obtained from the REOM to distinguish between 'mild' and 'very severe' COPD.
2. To collect descriptive information on the participant user experience with the REOM.
3. To determine concordance between the parameters obtained from the REOM and those obtained from the tremoflo oscillometry device with the 'standard' parameters obtained from each participant's standard Pulmonary Function Tests (PFT).

Hypothesis:

We hypothesize in the adult COPD patient population that the REOM parameter Reo1 and tremoflo device parameter R19 will correlate closely, and that the REOM parameter Reo2 and tremoflo device parameter R5 will correlate closely. We also hypothesize that the REOM, in particular, Reo2, will be able to distinguish between 'mild' and 'very severe' COPD, and that participants will report a positive user experience with the REOM.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged ≥40 with COPD, former/current smokers with a ≥10 pack-year smoking history.
* Diagnosed with COPD by FEV1/FVC < 0.7 using standard PFT post-bronchodilator testing, with either 'mild' ('GOLD 1': FEV1 ≥ 80% of predicted value) COPD or 'very severe' ('GOLD 4': FEV1 < 30% of predicted value) COPD.
* Ability to provide informed consent.

Exclusion Criteria:

* No existing COPD diagnosis
* History of co-morbid asthma
* Current use of home oxygen
* Any acute exacerbation of COPD (AECOPD) experienced within 4 weeks of participation in the study
* Chronic respiratory infection
* Any contraindication to respiratory testing
* Inability to participate in reproducible measurements due to physical or cognitive barrier

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with COPD at the Montreal Chest Institute (MCI) of the McGill University Health Centre (MUHC).
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-08-06 (Actual); Study Completion 2024-08-06 (Actual)

PRIMARY OUTCOMES:
Concordance (correlation) | Single-visit study: all tests performed at one single visit.
  Correlation will be tested using the Spearman correlation coefficient (r) between REOM-obtained (Reo1 and Reo2) and tremoflo-obtained (R19 and R5) resistance measurements.
Agreement | Single-visit study: all tests performed at one single visit.
  Agreement will be tested using the Bland-Altman test between REOM-obtained (Reo1 and Reo2) and tremoflo-obtained (R19 and R5) resistance measurements.

SECONDARY OUTCOMES:
Discriminative capacity | Single-visit study: all tests performed at one single visit.
  The t-test (between 2 independent means) will be used to determine the discriminative capacity of the REOM to distinguish between 'mild' and 'very severe' COPD.
Participant satisfaction and usability experience | Single-visit study: all tests performed at one single visit.
  Each participant will complete a 'participant satisfaction questionnaire' as well as the validated System Usability Scale (SUS) for each test (REOM, standard oscillometry, pulmonary function test). Data will be presented descriptively.

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No